CLINICAL TRIAL: NCT03140254
Title: A RANDOMIZED, SINGLE-CENTER, BLINDED, PILOT CLINICAL EVALUATION OF THE ANTIMICROBIAL EFFECTIVENESS OF THERMALLY TREATED CLOTHS IMPREGNATED WITH 0.4% OCTENIDINE DIHYDROCHLORIDE AQUEOUS SOLUTION COMPARED TO THERMALLY TREATED CLOTHS IMPREGNATED WITH VEHICLE FORMULATION AND TO SAGE 2% CHLORHEXIDINE GLUCONATE CLOTH FOR PREOPERATIVE SKIN PREPARATION
Brief Title: Evaluating Safety and Effectiveness of Octenidine Dihydrochloride
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MPS-16IPVAW01
Record Dates: First submitted 2016-09-19; First posted 2017-05-04 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Preoperative Skin Preparation
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- comparator (Active Comparator): Chlorhexidine gluconate
  Interventions: Drug: Chlorhexidine gluconate
- experimental (Experimental): BDIP-0001
  Interventions: Drug: N,N'-(1,10-decanediyldi-1(4H)-Pyridinyl-4-ylidene)-Bis-(1-octanamine) Dihydrochloride
- placebo (Placebo Comparator): Vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chlorhexidine gluconate
  Arms: comparator
Drug: N,N'-(1,10-decanediyldi-1(4H)-Pyridinyl-4-ylidene)-Bis-(1-octanamine) Dihydrochloride
  Arms: experimental
Drug: Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of a topical antiseptic for preoperative skin preparation

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of either sex, at least 18 years of age and of any race.
* Subjects must be in good general health.
* Subjects must read and sign an Informed Consent Form, Authorization to Use and Disclose Protected Health Information Form, and List of Restricted Products prior to participating in the study.
* Female subjects must have a negative urine pregnancy test documented before treatment with test materials.
* Screening day microbial baseline meeting minimum skin flora baseline requirements on abdomen and groin.

Exclusion Criteria:

* Known allergies or sensitivities to sunscreens, deodorants, laundry detergents, fragrances, vinyl, latex (rubber), alcohols, metals, inks, or to common antibacterial agents found in soaps, lotions, or ointments.
* Exposure of test sites to strong detergents, solvents, or other irritants within the 14-day product-restriction period or during the test period.
* Exposure of test sites to antimicrobial agents, medicated soaps, medicated shampoos, or medicated lotions, use of biocide-treated pools or hot tubs, use of tanning beds, or sunbathing during the 14-day product-restriction period or during the test period.
* Wear fabric softener-treated clothing (including bug-repellent and UV-treated clothing) during the 14-day product-restriction period or during the test period.
* Use of systemic or topical antibiotic medications, steroid medications (other than for hormonal contraception or post-menopausal reasons), or any other product known to affect the normal microbial flora of the skin during the 14-day product-restriction period or during the test period.
* A medical diagnosis of a physical condition, such as a current or recent severe illness, mitral valve prolapse with a heart murmur, congenital heart disease, hepatitis B, hepatitis C, an organ transplant, or an immunocompromised condition such as AIDS (or HIV positive), lupus, diabetes, Crohn's disease, asthma or medicated multiple sclerosis.
* Any tattoos, or scars within 2 inches of the test sites; skin blemishes or warts, may be permissible with the specific approval of the Principal Investigator or Consulting Physician.
* Dermatoses, cuts, lesions, active skin rashes, scabs, breaks in the skin or other skin disorders within 6 inches on or around the test sites.
* A currently active skin disease or inflammatory skin condition (for example, contact dermatitis, psoriasis, eczema) anywhere on the body that, in the opinion of the Principal Investigator, would compromise subject safety or study integrity.
* Subjects who receive an irritation score of 1 (any redness, swelling, rash, or dryness present at any treatment area) for any individual skin condition prior to the Screening Day baseline or Treatment Day baseline sample collection.
* Participation in another clinical study in the past 30 days or current participation in another clinical study.
* Showering, bathing, or swimming within the 72 hour period prior to sampling for baseline screening, the test day, or throughout the test period.
* Pregnancy, plans to become pregnant or impregnate a sexual partner within the pre-test and test periods of the study, or nursing a child. All female subjects will be required to complete a urine pregnancy test on the day of test material application, prior to treatment. Both gender of subjects must be willing to use an acceptable method of contraception to prevent pregnancy for at least 14 days immediately preceding Treatment Day and throughout the duration of the study.
* Any medical condition or use of any medications that, in the opinion of the Principal Investigator or Consulting Physician, would preclude participation.
* Unwillingness to fulfill the performance requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Burroughs, Study Director — Becton, Dickinson and Company
Locations (1):
- BioScience Laboratories, Butte, Montana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were only treated if they met baseline bacterial count criteria.
Groups:
- Treated Participants: Participants were treated with 2 of 3 study products, Investigational Product (IP, 0.4% OCT cloth), Vehicle Control (VC, vehicle formulation cloth), and/or Active Control (AC, SAGE 2% CHG cloth), 1 on the left side of the body (abdomen and inguen received the same product) and 1 on the right (abdomen and inguen received the same product). Therefore, treatment groups are not discrete categories and cannot be described by treatment group.
Period: Overall Study
Arm/Group | Treated Participants
Started | 145
Treatment IP - Groin | 51
Treatment IP - Abdomen | 48
Treatment AC - Groin | 51
Treatment AC - Abdomen | 48
Treatment VC - Groin | 18
Treatment VC - Abdomen | 19
Completed | 144
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Participants were treated with 2 of 3 study products, Investigational Product (IP, 0.4% OCT cloth), Vehicle Control (VC, vehicle formulation cloth), and/or Active Control (AC, SAGE 2% CHG cloth), 1 on the left side of the body (abdomen and inguen received the same product) and 1 on the right (abdomen and groin received the same product). Therefore, treatment groups are not discrete categories and cannot be described by treatment group.
Arm/Group | Treated Participants
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 132
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 124
  More than one race | 0
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Abdominal Site Responder Rates at 10 Minutes
Description: Individual anatomical sites were considered responders based on the standards set forth in the Food and Drug Administration Tentative Final Monograph for Effectiveness Testing of a Patient Preoperative Skin Preparation (FR 59:116, 17 June 94, pp. 31450-31452). Individually treated abdomen sites with a 2 log10/cm^2 CFU reduction were considered "responders," and individually treated groin sites with a 3 log10/cm^2 CFU reduction were considered "responders."
Time Frame: 10 min
Population: Number of individual sites that met treatment day bacterial requirements on the abdomen for analysis are IP = 48, AC = 48, VC = 19
Measure: Mean (95% Confidence Interval); unit: percentage of abdomen sites
Units Other Than Participants: Individual abdominal sites
Groups:
- Investigational Product: Investigational Product (IP) BDIP-0001
  N,N'-(1,10-decanediyldi-1(4H)-Pyridinyl-4-ylidene)-Bis-(1-octanamine) Dihydrochloride
- Active Control: Active Control (AC) Sage 2% Chlorhexidine gluconate
- Vehicle Control: Vehicle Control (VC)
Arm/Group | Investigational Product | Active Control | Vehicle Control
Number analyzed (Participants) | 77 | 81 | 34
Number analyzed (Individual abdominal sites) | 48 | 48 | 19
percentage of abdomen sites | 79.2 [65.7 to 88.3] | 85.4 [72.8 to 92.8] | 52.6 [31.7 to 72.7]

2. Primary Outcome: Percentage of Abdominal Site Responder Rates at 6 Hours
Description: Individual anatomical sites were considered responders based on the standards set forth in the Food and Drug Administration Tentative Final Monograph for Effectiveness Testing of a Patient Preoperative Skin Preparation (FR 59:116, 17 June 94, pp. 31450-31452). Individually treated abdomen sites with a log10/cm^2 CFU reduction greater than or equal to 0 were considered responders.
Time Frame: 6 hours
Population: Number of abdomen sites passing treatment day bacterial requirements were analyzed for responder rates. The number of anatomical sites meeting treatment day bacterial requirements were IP = 48, AC = 48, VC = 19 for the abdomen.
Measure: Mean (95% Confidence Interval); unit: percentage of abdomen sites
Units Other Than Participants: Individual Abdomen sites
Arm/Group | Investigational Product | Active Control | Vehicle Control
Number analyzed (Participants) | 77 | 81 | 34
Number analyzed (Individual Abdomen sites) | 48 | 48 | 19
percentage of abdomen sites | 89.6 [77.8 to 95.5] | 100.0 [92.6 to 100.0] | 94.7 [75.4 to 99.1]

3. Primary Outcome: Percentage of Groin Site Responder Rate at 6 Hours
Description: Individual anatomical sites were considered responders based on the standards set forth in the Food and Drug Administration Tentative Final Monograph for Effectiveness Testing of a Patient Preoperative Skin Preparation (FR 59:116, 17 June 94, pp. 31450-31452). Individually treated groin sites with a log10/cm^2 CFU reduction greater than or equal to 0 were considered responders.
Time Frame: 6 hours
Population: Individual sites that met treatment day bacterial requirements were analyzed for responder rates. Number of sites passing treatment day bacterial requirements on the groin were IP = 51, AC = 51, and VC = 18.
Measure: Mean (95% Confidence Interval); unit: percentage of groin sites
Units Other Than Participants: Individual Groin Sites
Arm/Group | Investigational Product | Active Control | Vehicle Control
Number analyzed (Participants) | 72 | 74 | 21
Number analyzed (Individual Groin Sites) | 51 | 51 | 18
percentage of groin sites | 100 [93 to 100] | 98 [89.7 to 99.7] | 100 [82.4 to 100]

4. Primary Outcome: Percentage of Groin Sites Responder Rates at 10 Minutes
Description: Participants were considered responders based on the standards set forth in the Food and Drug Administration Tentative Final Monograph for Effectiveness Testing of a Patient Preoperative Skin Preparation (FR 59:116, 17 June 94, pp. 31450-31452). Individually treated groin sites with a 3 log10/cm^2 CFU reduction were considered "responders."
Time Frame: 10 minutes
Population: Number of individually treated groin sites that passed treatment day bacterial requirements were IP = 51, AC = 51, and VC = 18.
Measure: Mean (95% Confidence Interval); unit: percentage of groin sites
Units Other Than Participants: Individual Groin Sites
Arm/Group | Investigational Product | Active Control | Vehicle Control
Number analyzed (Participants) | 73 | 74 | 21
Number analyzed (Individual Groin Sites) | 51 | 51 | 18
percentage of groin sites | 72.5 [59.1 to 82.9] | 74.5 [61.1 to 84.5] | 55.6 [33.7 to 75.4]

ADVERSE EVENTS:
Time Frame: 6 hours
Groups:
- All Participants: Participants were treated with 2 of 3 study products, Investigational Product (IP, 0.4% OCT cloth), Vehicle Control (VC, vehicle formulation cloth), and/or Active Control (AC, SAGE 2% CHG cloth), 1 on the left side of the body (abdomen and inguen received the same product) and 1 on the right (abdomen and inguen received the same product). Therefore, treatment groups are not discrete categories and cannot be described by treatment group.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/145
Serious Adverse Events (participants affected / at risk) | 0/145
Other Adverse Events (participants affected / at risk) | 0/145

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT03140254/Prot_SAP_000.pdf